CLINICAL TRIAL: NCT02133976
Title: Comparative Mechanisms (Mediators, Moderators) of Psychosocial Chronic Pain Treatments
Brief Title: Comparative Mechanisms of Psychosocial Chronic Pain Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Duke University (Other); University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12101001
Record Dates: First submitted 2014-05-05; First posted 2014-05-08 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; psychosocial interventions; mechanisms
MeSH Terms: interventions — Cognitive Behavioral Therapy; Behavior Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- cognitive therapy (Active Comparator): Cognitive therapy will be delivered to decrease pain interference
  Interventions: Behavioral: cognitive therapy; Other: treatment as usual
- mindfulness training (Active Comparator): Mindfulness training will be delivered to decrease pain interference
  Interventions: Behavioral: mindfulness training; Other: treatment as usual
- behavior therapy (Active Comparator): Behavior therapy will be delivered to decrease pain interference
  Interventions: Behavioral: behavioral therapy; Other: treatment as usual
- treatment as usual (Active Comparator): Subjects will engage in their usual care for low back pain.
  Interventions: Other: treatment as usual

INTERVENTIONS:
Behavioral: cognitive therapy
  Arms: cognitive therapy
Behavioral: mindfulness training
  Arms: mindfulness training
Behavioral: behavioral therapy
  Arms: behavior therapy
Other: treatment as usual

SUMMARY:
Psychosocial interventions are attractive options for treating chronic low back pain, and many approaches now have strong support for efficacy. However, few empirical data address whether psychosocial pain treatments work because of mechanisms specified by theory, and thus investigators know very little about HOW our treatments work. It may be that different treatments work via distinct pathways that are specific to a given treatment (single effect model), or it may be that different treatments work to the extent they all operate via key mechanisms that they share (additive effects model). Examination of specific and/or shared effects on outcomes of mechanisms will provide theoretical and empirical rationale for enhancing procedures and techniques most closely linked to strong outcomes and incorporating them into future interventions, while limiting the use of others that may be revealed as inert.

ELIGIBILITY:
Inclusion Criteria:

* significant daily chronic pain intensity (at least 4 on a 10-point scale; see below) and interference in performing daily activities due to pain (at least 3 on a 6-point scale; see below) for at least 6 months
* musculoskeletal pain of the low back and/or leg pain that may be related to history of degenerative disk disease, spinal stenosis, or disk herniation (radiculopathy subcategory), or muscular or ligamentous strain (chronic myofascial pain subcategory)
* age between 18 and 75 years.

Exclusion Criteria:

* meet criteria for alcohol or substance abuse problems
* meet criteria for past or present psychotic or bipolar disorders
* inability to understand English well enough to complete questionnaires or to participate in therapy
* active suicidal ideation with intent
* pain is due to malignant conditions (eg, cancer, rheumatoid arthritis), migraine or tension headache, fibromyalgia or complex regional pain syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Pain interference | 12 months
  Pain interference will be assessed with Pain Interference Subscale items of the Multidimensional Pain Inventory

SECONDARY OUTCOMES:
Activity level | 12 months
  Activity level will be assessed with the General Activity subscale items of the Multidimensional Pain Inventory, and via actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: John W Burns, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Gerhart J, Burns JW, Thorn B, Jensen M, Carmody J, Keefe F. Treatment mechanism and outcome decoupling effects in cognitive therapy, mindfulness-based stress reduction, and behavior therapy for chronic pain. Pain. 2025 Feb 1;166(2):408-419. doi: 10.1097/j.pain.0000000000003374. Epub 2024 Aug 30. PMID 39226076
- [Derived] Burns JW, Jensen MP, Thorn BE, Lillis TA, Carmody J, Gerhart J, Keefe F. Cognitive Therapy, Mindfulness-Based Stress Reduction, and Behavior Therapy for the Treatment of Chronic Pain: Predictors and Moderators of Treatment Response. J Pain. 2024 Jun;25(6):104460. doi: 10.1016/j.jpain.2024.01.003. Epub 2024 Jan 8. PMID 38199593
- [Derived] Burns JW, Jensen MP, Gerhart J, Thorn BE, Lillis TA, Carmody J, Keefe F. Cognitive therapy, mindfulness-based stress reduction, and behavior therapy for people with chronic low back pain: A comparative mechanisms study. J Consult Clin Psychol. 2023 Mar;91(3):171-187. doi: 10.1037/ccp0000801. Epub 2023 Feb 27. PMID 36848061
- [Derived] Burns JW, Jensen MP, Thorn B, Lillis TA, Carmody J, Newman AK, Keefe F. Cognitive therapy, mindfulness-based stress reduction, and behavior therapy for the treatment of chronic pain: randomized controlled trial. Pain. 2022 Feb 1;163(2):376-389. doi: 10.1097/j.pain.0000000000002357. PMID 34074945